CLINICAL TRIAL: NCT00560729
Title: Effectiveness and Cost of a Quantitative and Qualitative Nutritional Supplementation in Elderly Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCNF 0402
Record Dates: First submitted 2007-11-06; First posted 2007-11-20 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Denutrition
Keywords: elderly people

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- I (No Intervention)
- II (Active Comparator): oral nutrition
  Interventions: Dietary Supplement: Renutryl 500
- III (Experimental): oral nutrition
  Interventions: Dietary Supplement: Generique
- IV (Experimental): oral nutrition
  Interventions: Dietary Supplement: Generique + Renutryl 500

INTERVENTIONS:
Dietary Supplement: Renutryl 500
  Arms: II
Dietary Supplement: Generique
  Arms: III
Dietary Supplement: Generique + Renutryl 500
  Arms: IV

SUMMARY:
Evaluation of the effectiveness and the costs of a quantitative and qualitative nutritional supplementation in elderly patients

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization into a geriatric care unit
* age > 70 years
* C reactive protein > 30 mg/l
* 25 < albumin < 35 g/l
* 130 < Na < 145 mmol/l
* BMI < 22
* weight loss > 10 % within the last 6 months
* MNA < 23.5

Exclusion Criteria:

* diabetes mellitus
* severe digestive failure
* enteral or parenteral nutrition
* renal,cardiac or digestive failure
* lactose intolerance
* terminal phase severe pathology
* MMS < 15

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 63 (Actual)
Dates: Start 2003-10; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Nutritional Risk Index | At J0, J21, J42

SECONDARY OUTCOMES:
Measure of body mass index (BMI), Mini Nutritional Assessment, Fat mass,lean mass, serum albumin and transthyretin,Activities of Daily Living (ADL), ingesta and morbidity.
Tolerance | Daily

CONTACTS AND LOCATIONS:
Overall Officials: Christian Aussel, PhD, Study Director — University PARIS V
Locations (3):
- France (3):
  - Hôpital Georges Clemenceau, Champcueil
  - Hopital Emile Roux, Limeil-Brévannes
  - Hopital Charles RICHET, Villiers-le-Bel